CLINICAL TRIAL: NCT03275025
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Therapeutic Exploratory, Phase II Clinical Trial for the Efficacy Investigation and Safety Evaluation of YRA-1909 in Patients With Rheumatoid Arthritis Who Are on a Stable Dose of Methotrexate (MTX) and Who Have an Inadequate Response to MTX (MTX-IR)
Brief Title: A Phase 2 Study to Evaluate the Safety and Efficacy of YRA-1909 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yungjin Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YJ15-201
Record Dates: First submitted 2017-08-28; First posted 2017-09-07 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- YRA-1909 low dose (Experimental)
  Interventions: Drug: YRA-1909 low dose; Drug: Placebo
- YRA-1909 medium does (Experimental)
  Interventions: Drug: YRA-1909 mid dose; Drug: Placebo
- YRA-1909 high dose (Experimental)
  Interventions: Drug: YRA-1909 high dose
- YRA-1909 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YRA-1909 low dose — A low dose of YRA-1909; daily oral intake for 12 weeks
  Arms: YRA-1909 low dose
Drug: YRA-1909 mid dose — A mid dose of YRA-1909; daily oral intake for 12 weeks
  Arms: YRA-1909 medium does
Drug: YRA-1909 high dose — A high dose of YRA-1909; daily oral intake for 12 weeks
  Arms: YRA-1909 high dose
Drug: Placebo — Matching placebo dosing with daily oral intake for 12 weeks
  Arms: YRA-1909 Placebo; YRA-1909 low dose; YRA-1909 medium does

SUMMARY:
This is a multicenter, randomized, double-blind phase2 study to evaluate the safety and investigate the efficacy of YRA-1909 in Patients with Rheumatoid Arthritis who are on a stable dose of Methotrexate(MTX) and who have an inadequate response to MTX(MTX-IR).

ELIGIBILITY:
Inclusion Criteria:

* 19 Years to 80 Years
* Subjects with onset RA classified by ACR/EULAR 2010 revised classification criteria at least 12 weeks prior to screening
* Subjects meet the ACR 1992 Revised Criteria for the Classification of Global Functional Status in RA Class I, II or, III at screening

Exclusion Criteria:

* Subjects meet the ACR 1992 Revised Criteria for the Classification of Global Functional Status in RA Class Ⅳ at screening
* Any of the following laboratory values at screening:

  1. Patients with severe liver impairment (AST or ALT > 2 times the upper limit of normal)
  2. Patients with renal disease,immunodeficiency disease and peptic ulcer
  3. Patients with pleural effusion and ascites

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
American College of Rheumatology 20 (ACR20) response rate at Week 12 | Week 12
Percentage of Participants With Adverse Events | Week 12
  Incidence of all grade adverse events

SECONDARY OUTCOMES:
ACR20 Response at Week 4,8 | Week 4 and 8
Change From Baseline in Patient Assessment of Pain Visual Analog Scale (VAS) at Week 4,8 and 12 | Week 4,8 and 12
ACR 50, 70 Response at Week 4, 8 and 12 | Week 4, 8 and 12
Mean Percent Change From Baseline in the Swollen Joint Count(SJC) and Tender Joint Count (TJC) at Week 4, 8 and 12 | Week 4, 8 and 12
Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Week 4, 8 and 12 | Week 4, 8 and 12
Change From Baseline in High Sensitivity C-Reactive Protein (hsCRP) at Week 4, 8 and 12 | Weeks 4, 8 and 12
Mean Change from Baseline in Assessment of participant's illness at Week 4, 8 and 12 by participants and investigator/sub-investigator | Week 4, 8 and 12

CONTACTS AND LOCATIONS:
Overall Officials: YeongWook Song, M.D.,Ph.D., Study Chair — Seoul National University Hospital
Locations (14):
- South Korea (14):
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Hanllym University Medical Center, Anyang
  - Chungbuk National University Hospital, Chungju
  - Kelmyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Kyung Hee University Hospital at Gangdong, Gangdong
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam
  - Hanyang University Seoul Hospital, Seoul
  - KyungHee University Hospital, Seoul
  - Seoul Metropolitan Goverment Seoul National Univeersity Boramae Medical Center, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No